CLINICAL TRIAL: NCT06272890
Title: The Effect of Motivational Interviewing on Social Anxiety Level, Dating Violence and Self-compassion in Nursing Students With Social Anxiety: a Randomized Controlled Study
Brief Title: The Effect of Motivational Interviewing on Nursing Students
Acronym: mg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Merve Işık, Asst.Prof.Dr., Giresun University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GiresunU
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Motivation
Keywords: social anxiety; nursing students; dating violence; motivational interview; self-compassion
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: The research was planned as a randomized controlled experimental study in a two-center parallel group pretest-posttest design.
Who Masked: Outcomes Assessor
Masking Description: In order to prevent detection bias in the study, all measurements will be made using an online survey form. In order to prevent reporting bias, the data obtained from the research will be coded as A and B by an independent statistician, transferred to the SPSS program and analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group will receive online motivational interviewing (MI) consisting of five sessions. The sessions are planned to take place on the same day and time every week. Each session will last an average of 40 minutes. In the literature, PD sessions with groups of 5-8 people have been evaluated as adequate and effective. Before the MG, a WhatsApp group will be established to provide faster and easier communication to the intervention group and communication about the sessions will be handled in this group.
  Interventions: Behavioral: motivational interviewing
- control group (No Intervention): No treatment will be applied to the control group during the study period.

INTERVENTIONS:
Behavioral: motivational interviewing — motivational interviewing
  Arms: intervention group

SUMMARY:
Studies support the idea that people diagnosed with social anxiety disorder score significantly lower on self-acceptance than healthy controls, and that self-compassion is inversely related to anxiety. Motivational interviewing has been shown to improve treatment outcomes as well as predict higher self-compassion and reduced resistance among participants.It also has the ability to increase the effectiveness of motivational interviewing as an intervention with perpetrators of intimate partner violence, promoting readiness for change and progression through stages of change. In this context, this study aims to examine the effect of motivational interviewing on social anxiety level, dating violence and self-compassion in nursing students with social anxiety.

DETAILED DESCRIPTION:
Nursing as a social profession needs more social interaction. Nurses should be able to develop therapeutic interaction with patients. This can only be possible when they are confident in themselves and worry about others and get rid of anxiety disorders. Social anxiety symptoms have been associated with increased risk of depression, other anxiety disorders and substance misuse, as well as difficulties in making healthy social connections and adjusting to the academic environment. Motivational interviewing (MI) has been found to provide symptom reduction in individuals with generalized anxiety disorder and to improve treatment outcome in individuals with SAD. A meta-analysis by Kirby et al. (2017) concluded that existing self-compassion-based interventions are moderately successful in enhancing compassion and reducing suffering (e.g. depression, anxiety, distress). While moderate effects are very important and encouraging, they indicate that interventions can be improved. It is suggested that including PD as a prelude to compassion-based interventions may provide similar benefits for program participation, initiation, adherence, and behavior change.It has also been shown that PD may increase sensitivity to dating violence interventions. In this context, this study aims to examine the effect of motivational interviewing on social anxiety level, dating violence and self-compassion in nursing students with social anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Have moderate and severe social anxiety (55 and above LSCQ)
* Volunteering to participate in the research
* Being in the pre-intention and intention stage according to the stage of change assessment form

Exclusion Criteria:

* Have to no or low level of social anxiety (below of 55 on the LSCQ)
* Have to any psychiatric diagnosis
* Have received psychotherapy for social anxiety before
* Attend to a psychotherapy or counseling program

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2024-04-20 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Motivational interviewing has an effect on nursing students' social anxiety. | Change from before implementation and 5th week of the practice

SECONDARY OUTCOMES:
Motivational interviewing has an effect on nursing students' dating violence. | Change from before implementation and 5th week of the practice

OTHER OUTCOMES:
Motivational interviewing has an effect on nursing students' self-compassion. | Change from before implementation and 5th week of the practice

CONTACTS AND LOCATIONS:
Overall Officials: Sultan Özkan Şat, PhD, Principal Investigator — Bitlis Eren University; Pınar Akbaş, PhD, Principal Investigator — Karabük University
Locations (1):
- Giresun University, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided